CLINICAL TRIAL: NCT06662916
Title: Microbiota-Diversity Enhancing Diet on Children With Autism Spectrum Disorder: The MIND-DASE Study
Brief Title: Gut Microbiota Diversity: Wrong Message in Autism, Wrong Architecture in Formation
Status: Completed | Type: Observational
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Hasan Onal, MD, Prof M.D., Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: SBUCAMSAKURAEAH
Record Dates: First submitted 2024-10-17; First posted 2024-10-29 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Autism Spectrum Disorder; Gut -Microbiota; Neurodevelopment Outcome
Keywords: Autism Spectrum Disorder; Microbiota Diversity; Diet; Neurodevelopment outcome
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 220 ASD cases regularly followed our specific diet: 220 individuals who regularly followed our specific diet program for at least 12 months were identified as a study group.
  Interventions: Behavioral: Microbiota-Diversity Enhancing Diet on children with Autism Spectrum Disorder
- 100 ASD cases who did not have diet compliance: 100 children with ASD who did not have diet compliance were identified as control group.

INTERVENTIONS:
Behavioral: Microbiota-Diversity Enhancing Diet on children with Autism Spectrum Disorder — Microbiota-Diversity Enhancing Diet on Children with ASD (MIND-DASE) suggested that increasing microbiota diversity through dietary interventions can have significant benefits on the neurodevelopmental outcomes of children with ASD
  Groups: 220 ASD cases regularly followed our specific diet

SUMMARY:
Our dietary diversity has changed day by day in industrial age. A low dietary diversity may alter gut microbiota diversity and functional capacity. Wrong messages sourced from gut microbiota were speculated to have a bad influence on autism spectrum disorder (ASD) severity. A new nutritional model aiming to increase microbiota diversity in children with ASD can improve social and communicative behaviors in these children. The investigators compared 220 ASD patients who regularly followed a specific diet program for at least 12 months with randomly selected 100 children with ASD who did not have diet compliance in terms of nutritional status and regular behavioral assessments with special scales (ATEC, ABC, QoLA-P scales). The investigators arised a question that the Microbiota-Diversity Enhancing Diet on Children with ASD (MIND-DASE) which is a specific dietary intervention may have benefits on the neurodevelopmental outcomes of children with ASD.

DETAILED DESCRIPTION:
Since industrialization has altered human diet models, we faced with a low dietary diversity, reduced gut microbiota diversity and functional capacity day by day. These changes in gut microbiota have been speculated to associate with severity of autism spectrum disorder (ASD). The investigators researched the possible therapeutic effects of a new nutritional model aiming to increase microbiota diversity in children with ASD. Question is: Can we improve social and communicative behaviors in children with ASD by increasing microbiota diversity through a specific diet? A total of 2000 children diagnosed with ASD and followed in Autism Nutrition Research Center in investigators' hospital were screened: a) a total of 220 participants aged between 2-18 years who regularly followed the specific diet program for at least 12 months were identified as a study group, and b) randomly selected 100 children with ASD who did not have diet compliance were identified as control group. Assessments included dietary adherence and behavioral evaluations using baseline, 6th and 12th month Autism Treatment and Evaluation Checklist (ATEC), Aberrant Behavior Checklist (ABC), The Quality of Life in Autism Questionnaire- Parent version (QoLA-P) scales. The investigators compared diet and non-diet groups by evaluating demographic data, clinical symptoms, diet compliance status and ATEC, ABC, and QoLA-P scores in 12-month time period. The investigators foced on The Microbiota-Diversity Enhancing Diet on Children with ASD (MIND-DASE) which is a specific dietary intervention may have significant benefits on the neurodevelopmental outcomes of children with ASD.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who were diagnosed ASD by a pediatric psychiatrist or a pediatric neurologist according to the DSM-V criteria
* Having continued follow-up in our center at least 12 months regularly
* Being between the ages of 2-18

Exclusion Criteria:

* Having a genetic syndrome (such as Rett, Angelman syndrome)
* Having an additional chronic disease
* Following a different diet program other than our center

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 320 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Changes in ATEC scores in diet (study) and non-diet (control) ASD participants from baseline to 1 year period. | From enrollment to the end of 12-month time period
  ATEC scores will be evaluated by a specialist psychiatric nurse in both groups. ATEC is a parent-completed questionnaire and has four subscales. A total score, which ranges from 0-179 points, is calculated from combined scores of each subscale. A lower ATEC score indicates improvement of ASD symptoms and a higher score correlates with more severe symptoms.
Changes in ABC scores in diet (study) and non-diet (control) ASD participants from baseline to 1 year period. | From enrollment to the end of 12-month time period
  ABC scores will be evaluated by a specialist psychiatric nurse in both groups. ABC is a scale for determining the behavioral problems in ASD children. It consists of 5 subscales and 58 items. Each item is rated on a four-point scale ranging from 0 (not a problem) to 3 (the problem is severe). Evaluation is based on the scores obtained from the subscales; minimum 0 points to maximum 174 points.
Changes QoLA-P scores in diet (study) and non-diet (control) ASD participants from baseline to 1 year period. | From enrollment to the end of 12-month time period
  The QoLA-P scores will be evaluated by a specialist psychiatric nurse in both groups.
  QoLA-P is designed as two subscales: Section A evaluates parent's perceptions about their own QoL, and section B measures the perceptions of parent's problems lived with an autistic child. Total score from this questionnaire ranges from 48 to 240 and higher scores show lesser severity effect.

SECONDARY OUTCOMES:
Height status in diet and non-diet group | From enrollment to the end of 12-month time period
  Participants' height (cm) values will be recorded at baseline and 3-month intervals. These values will be compared in between the groups during the time period.
Weight status in diet and non-diet group | From enrollment to the end of 12-month time period
  Participants' weight (kg) values will be recorded at baseline and 3-month intervals. These values will be compared in between the groups during the time period.

OTHER OUTCOMES:
Observation of eating pattern | From enrollment to the end of 12-month time period
  A selective eating pattern such as food rejection, food selectivity, excessive and persistent consumption of selected food will be recorded in the participants. The rate of diet compliance will be determined in ASD patients. We will observe whether these families have difficulty in adapting to the diet.

CONTACTS AND LOCATIONS:
Locations (1):
- Basakşehir Cam & Sakura City Hospital, Autism Nutrition and Research Center, Istanbul, Basaksehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes